CLINICAL TRIAL: NCT04768621
Title: Health Consequences of Wintering in the French Southern and Antarctic Territories
Acronym: MediTAAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020/CHU/38
Record Dates: First submitted 2021-02-17; First posted 2021-02-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2021-02

CONDITIONS: Environmental Exposure; Winter Depression; Endocrine System Diseases; Sleep Disorder; Immunologic Activity Alteration
MeSH Terms: conditions — Seasonal Affective Disorder; Endocrine System Diseases; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Winter residents of Southern and Antartic French Lands, (Experimental): people exposed to stressors over long periods including winter
  Interventions: Other: Questionary
- Country people going to Southern and Antartic French Lands (Active Comparator): people going to Southern and Antarctic French Lands who benefit from milder conditions and only make short stays
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — Questions about patient health after wintering in Southern and Antarctic French Lands about social and demographics items, psychologic and psychiatric items, sleep disorders, immunological disorders,and endocrinologic disorders, sociological consequences of wintering

SUMMARY:
Polar stays expose people to extreme climate, isolation and confinement. The combination of these factors induces psychological disorders, sleep disorders, immune and endocrine disturbances, and deficiencies. In the TAAF, (French Southern and Antarctic Lands) two types of population coexist: winter residents, exposed to these stressors over long periods, and country people, who benefit from milder conditions and only make short stays. In this context, the investigators have decided to set up this cohort study with the objective of comparing the state of health of the winterers of the TAAF from 2012 to 2017 with that of the country people of the same period, before their stay, during and the year following their return.

DETAILED DESCRIPTION:
Participants will answer to a questionnaire. This questionnaire will determinate participants health about following areas : psychological disorders, sleep disorders, immune and endocrine disturbances, and any deficiencies.

ELIGIBILITY:
Inclusion Criteria:

for the exposed group are:

* To have carried out one or more wintering in one of the districts of the TAAF, that means a stay of at least six consecutive months including winter;
* Have started their first wintering between 01jan2012 and 31dec2017;
* Know how to read and write French.

for the non-exposed group are:

* To have taken part in one or more summer campaigns between 01jan2012 and 31dec2017;
* Never have overwintered;
* Not having been refused wintering for health reasons or following psychological tests;
* Knowing how to read and write French.

Exclusion Criteria:

* Persons under guardianship or guardianship, deceased persons, persons refusing to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Evaluate incidence health disorders and sociological consequences of wintering of health of winterers (exposed) of TAAF from 2012 to 2017 with that of country people (not exposed) of the same period | between 4 years and 9 years after polar exposure
  Measurement tool is a questionnaire Prevalence of different pathologies will be described
  * Sociodemographic data
  * Psychological and psychiatric evaluation: Psychiatric disorder according to the College of Psychiatry Teacher; Assessment of coping strategy according to the Ways of Coping Checklist, a psychometric assessment tool recognized in the social science
  * Subjective perception of the state of health
  * Sleep disorder according to the definition of the College of Teacher of Neurology
  * Immunological state through the exploration of allergy according to College of Pulmonology Teacher, autoimmune disease according to the French College of Rhumatology Teacher (COFER), and infection by using the classification of infectious disease as presented in the Inserm epidemiological report
  * Endocrine pathology: dysthyroidism, vitamin D deficiency assessed by its complication as described by COFER
  * other pathologies presented in International Classification Disease

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOUSCAREN, Principal Investigator — CIC 1410
Locations (1):
- CHU de la Réunion, Saint-Denis, Reunion